CLINICAL TRIAL: NCT00199368
Title: A Long-Term, Multicenter, Open-Label Safety Study With Oral 20 or 40 mg/d Doses of KW-6002 (Istradefylline) as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa Therapy.
Brief Title: An Extension of Istradefylline in Parkinson's Disease Patients Who Have Completed Studies 6002-EU-007, 6002-US-013 or 6002-US-018
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6002-INT-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline ( KW-6002)

SUMMARY:
This is a 1-year, open-label, long-term safety extension for patients who have completed prior istradefylline studies 6002-EU-007, 6002-US-013 or 6002-US-018.

DETAILED DESCRIPTION:
Patients with Parkinson's disease with motor complications on levodopa therapy who completed the prior double-blind studies 6002-EU-007, 6002-US-013 or 6002-US-018 are eligible to enter into this 1-year, long-term open safety study with a starting istradefylline dose of 40mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study 6002-EU-007, 6002-US-013 or 6002-US-018
* Non-pregnant and either not of childbearing potential or using specified contraception

Exclusion Criteria:

* History of psychotic illness
* Variant/atypical Parkinson's disease
* Cancer within 5 years of enrollment
* ALT/AST levels > 1.5 times ULN
* Seizure disorder
* Neuroleptic malignant syndrome

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2004-10; Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Kyowa Pharmaceutical Inc., Princeton, New Jersey, United States